CLINICAL TRIAL: NCT04621448
Title: Extending Independence and Quality of Life for People With Alzheimer's Disease or Dementia Through Telehealth Program Delivery
Brief Title: Moving Together: An Online Group Movement Program for People Living With Memory Loss and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: R44AG059520 (NIH); R44AG059520 (NIH)
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Delayed-start control group
Who Masked: Outcomes Assessor
Masking Description: Dyads will be enrolled and randomized in blocks of 16 (n=8 immediate start, n=8 waitlist). The randomization sequence will be generated in advance by Dr. Barnes' team using a random number generator and will be maintained in a secure location. Individuals who collect or analyze outcome data will be unaware of the randomization sequence and blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Start (Experimental): The Immediate Start group will participate in the 12-week Moving Together program after completing the baseline assessment. Moving Together is a gentle, live-streaming, group movement program designed specifically for people with memory loss (PWML) and caregivers (CG) to do together. It is based on the in-person Preventing Loss of Independence through Exercise (PLIÉ) and Paired PLIÉ programs. The program combines physical movements to help maintain daily function with mindful body awareness exercises and social interactions to provide a comprehensive, multi-domain program.
  Interventions: Behavioral: Moving Together
- Delayed Start (Experimental): A Delayed Start group will be encouraged to continue with their usual daily activities during the first 12 weeks of the study and will begin the Moving Together program after completing the mid-point assessment.
  Interventions: Behavioral: Moving Together

INTERVENTIONS:
Behavioral: Moving Together — Two-way livestreaming virtual group classes will be offered for 1 hour, 2 days/week for 12 weeks to all participants. Classes will be led by a trained instructor who will demonstrate all movements and will provide brief explanations for the goals of movements. Consistent with the in-person program, classes will focus on the 7 guiding principles of Moving Together:
  1. repetition with variation (to promote procedural learning);
  2. progressive, functional movements (to improve daily function);
  3. slow pace and step-by-step instruction (to minimize cognitive demands);
  4. participant-centered goal orientation (to enhance personal meaningfulness of movements);
  5. body awareness, mindfulness and breathing (to encourage present-centeredness);
  6. social interaction (to promote meaningful connection); and
  7. positive emotions (to promote feelings of well-being.
  Other Names: Together Senior Health

SUMMARY:
To determine whether Moving Together improves quality of life in people with memory loss (PWML) and caregivers (CG) by performing a randomized, controlled trial (RCT) with a waitlist control group in 224 dyads.

DETAILED DESCRIPTION:
The investigators will perform an RCT with a 12-week delayed start control group in 224 dyads of PWMLs and CGs. The primary outcome in PWML will be self-rated quality of life (Quality of Life in Alzheimer's Disease, QOL-AD). Secondary outcomes will include: a) self-reported emotional well-being; b) self-reported social isolation; c) self-reported mobility; and d) directly assess cognitive performance. In CGs, the primary outcome will be self-rated quality of life (SF-12). Secondary outcomes in CGs will include: a) healthy days; b) self-efficacy; c) burden; d) social isolation; e) ability to self-regulate; f) positive affect; and g) sleep quality. In addition, the investigators will ask CGs to report sleep quality, mobility, and cognitive function for PWML. Additional exploratory outcomes will include health services utilization (hospitalizations, emergency department visits) and falls.

In addition to the RCT, the investigators propose to compare health utilization outcomes in study participants to a matched 'no contact' comparison sample of patients with dementia diagnoses who receive care in the University of California San Francisco (UCSF) Health system.

ELIGIBILITY:
Inclusion Criteria:

* People with memory loss (PWML):

  * U.S. resident;
  * English language fluency;
  * diagnosis of Alzheimer's disease or other dementia; mild severity, assessed using the Quick Dementia Rating System.
* Caregivers (CG):

  * U.S. resident;
  * English language fluency;
  * Primary caregiver for PWML;
  * own one or more devices that can be used to participate in two-way livestreaming video classes (e.g., smart phone/tablet + TV, laptop or desktop with webcam, smart TV);
  * willing and able to participate in two-way livestreaming group movement classes with person with PWML.

Exclusion Criteria:

* Age < 18 years;
* primarily use wheelchair inside home;
* limited life expectancy (e.g., enrolled in hospice, meta-static cancer);
* physical limitations that could affect ability to participate (e.g., difficulty sitting for 1 hour, chronic pain, vertigo);
* severe visual impairment (e.g., unable to observe instructor's movements on screen);
* severe hearing impairment (e.g., unable to hear instructor's requests);
* behavioral or psychiatric issues that could be disruptive in group setting (e.g., history of physical or verbal abuse, schizophrenia, bipolar disorder, substance abuse);
* unable to provide consent/assent;
* planning to travel for >1 week during initial 12-week study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Barnes, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Sharing permissions will be configured to ensure files containing PHI can only be accessed by authorized individuals. Two-step verification will be used as an additional safeguard against unauthorized access. Permissions will be updated when personnel roles change and they no longer need access to PHI or when they leave the research team.

REFERENCES:
- [Background] Barnes DE, Mehling W, Wu E, Beristianos M, Yaffe K, Skultety K, Chesney MA. Preventing loss of independence through exercise (PLIE): a pilot clinical trial in older adults with dementia. PLoS One. 2015 Feb 11;10(2):e0113367. doi: 10.1371/journal.pone.0113367. eCollection 2015. PMID 25671576
- [Background] Casey JJ, Harrison KL, Ventura MI, Mehling W, Barnes DE. An integrative group movement program for people with dementia and care partners together (Paired PLIE): initial process evaluation. Aging Ment Health. 2020 Jun;24(6):971-977. doi: 10.1080/13607863.2018.1553142. Epub 2019 Feb 12. PMID 30744387
- [Background] Wu E, Barnes DE, Ackerman SL, Lee J, Chesney M, Mehling WE. Preventing Loss of Independence through Exercise (PLIE): qualitative analysis of a clinical trial in older adults with dementia. Aging Ment Health. 2015;19(4):353-62. doi: 10.1080/13607863.2014.935290. Epub 2014 Jul 14. PMID 25022459
- [Background] Nicosia FM, Lee JA, Chesney MA, Benjamin C, Lee AN, Mehling W, Sudore RL, Barnes DE. Adaptation of an In-Person Mind-Body Movement Program for People with Cognitive Impairment or Dementia and Care Partners for Online Delivery: Feasibility, Satisfaction and Participant-Reported Outcomes. Glob Adv Integr Med Health. 2023 Sep 21;12:27536130231202989. doi: 10.1177/27536130231202989. eCollection 2023 Jan-Dec. PMID 37745819
- [Result] Barnes DE, Jiang F, Benjamin C, Lee JA, Sudore RL, Mehling WE, Chesney MA, Chao LL, Nicosia FM. Livestream, group movement program for people living with cognitive impairment and care partners: A randomized clinical trial. Alzheimers Dement (N Y). 2024 May 2;10(2):e12467. doi: 10.1002/trc2.12467. eCollection 2024 Apr-Jun. PMID 38698931
- See also: Published results — https://pmc.ncbi.nlm.nih.gov/articles/PMC11064212/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants are enrolled as dyads of persons living with dementia (PLWD) and care partners (CPs).
Groups:
- Waitlist Control - PLWD: Usual activities for 12 weeks followed by Moving Together classes (1 hour, 2 days/week) for 12 weeks for PLWD.
- Moving Together - PLWD: Synchronous, online, mind-body group movement classes (1 hour, 2 days/week) for 12 weeks followed by optional continuation of classes for 12 weeks for PLWD.
- Waitlist Control - CP: Usual activities for 12 weeks followed by Moving Together classes for 12 weeks (1 hour, 2 days/week) for CPs.
- Moving Together - CP: Synchronous, online, mind-body group movement classes (1 hour, 2 days/week) for 12 weeks followed by optional continuation of classes for 12 weeks for CPs.
Period: Baseline to 12 Weeks
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD | Waitlist Control - CP | Moving Together - CP
Started | 43 | 54 | 43 | 54
Completed | 37 | 45 | 37 | 45
Not Completed | 6 | 9 | 6 | 9
Not completed — Withdrawal by Subject | 6 | 8 | 6 | 8
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Period: 12 to 24 Weeks
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD | Waitlist Control - CP | Moving Together - CP
Started | 37 | 45 | 37 | 45
Completed | 33 | 43 | 33 | 43
Not Completed | 4 | 2 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Participants enrolled as dyads of persons living with dementia (PLWD) and care partners (CPs).
Groups:
- Waitlist Control: Usual activities for 12 weeks followed by Moving Together classes (1 hour, 2 days/week) for 12 weeks.
- Moving Together: Synchronous, online, mind-body group movement classes (1 hour, 2 days/week) for 12 weeks followed by return to usual activities for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Waitlist Control | Moving Together | Total
Number analyzed (Participants) | 86 | 108 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There are separate rows for PLWD and CPs.
  years
    Participants with dementia: number analyzed (Participants) | 43 | 54 | 97
    Participants with dementia | 76.8 (9.7) | 76.2 (11.3) | 76.4 (10.6)
    Care partners: number analyzed (Participants) | 43 | 54 | 97
    Care partners | 68.9 (11.0) | 63.3 (11.8) | 65.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There are separate rows for PLWD and CPs.
  Participants
    Participants with dementia: number analyzed (Participants) | 43 | 54 | 97
    Participants with dementia: Female | 21 | 21 | 42
    Participants with dementia: Male | 22 | 33 | 55
    Care partners: number analyzed (Participants) | 43 | 54 | 97
    Care partners: Female | 32 | 44 | 76
    Care partners: Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: There are separate rows for PLWD and CPs.
  Participants
    Participants with dementia: number analyzed (Participants) | 43 | 54 | 97
    Participants with dementia: Asian | 3 | 5 | 8
    Participants with dementia: Black or African American | 1 | 4 | 5
    Participants with dementia: Hispanic/Latino/a/x (any race) | 2 | 1 | 3
    Participants with dementia: Non-Hispanic White | 36 | 42 | 78
    Participants with dementia: Other/unknown race/ethnicity | 1 | 2 | 3
    Care partners: number analyzed (Participants) | 43 | 54 | 97
    Care partners: Asian | 5 | 9 | 14
    Care partners: Black or African American | 0 | 5 | 5
    Care partners: Hispanic/Latino/a/x (any race) | 4 | 1 | 5
    Care partners: Non-Hispanic White | 33 | 36 | 69
    Care partners: Other/unknown race/ethnicity | 1 | 3 | 4
Education [Mean (Standard Deviation); unit: years] — Population: Separate rows are provided for PLWD and CPs
  years
    Participants with dementia: number analyzed (Participants) | 43 | 54 | 97
    Participants with dementia | 16.2 (3.1) | 16.8 (2.8) | 16.5 (3.0)
    Care partners: number analyzed (Participants) | 43 | 54 | 97
    Care partners | 17.0 (3.2) | 16.7 (2.8) | 16.8 (3.0)
Dementia Diagnosis [Count of Participants; unit: Participants] — Population: Measure only collected for PLWD
  Participants
    number analyzed (Participants) | 43 | 54 | 97
    Alzheimer's disease | 12 | 17 | 29
    Dementia unspecified | 4 | 15 | 19
    Mild cognitive impairment | 7 | 6 | 13
    Mixed dementia | 4 | 1 | 5
    Vascular dementia | 5 | 5 | 10
    Other/unknown type of dementia | 11 | 10 | 21
Quick Dementia Rating System (QDRS) [Mean (Standard Deviation); unit: points on a scale] — 10-item validated questionnaire. Scores range from 0 to 30 with higher scores indicating greater cognitive impairment. Enrollment restricted to participants with scores of 2.5 to 12.5 (mild severity). Population: Measure only relevant for PLWD.
  points on a scale
    number analyzed (Participants) | 43 | 54 | 97
    (all) | 7.5 (2.9) | 7.8 (2.3) | 7.7 (3.0)
Relationship to PLWD [Count of Participants; unit: Participants] — Population: Only relevant for CPs
  Participants
    number analyzed (Participants) | 43 | 54 | 97
    Spouse or partner | 31 | 34 | 65
    Child or child-in-law | 9 | 15 | 24
    Paid | 1 | 3 | 4
    Other relationship | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life - Change (Quality of Life in Alzheimer's Disease Scale, QOL-AD)
Description: The QOL-AD is a standard quality of life measure that has been validated for people with cognitive impairment. Scores may range from 0-52, with higher scores reflecting better quality of life.
Time Frame: Baseline to 12-weeks
Population: Only measured in PLWD. Baseline data missing for 1 participant in the Moving Together group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Waitlist Control - PLWD: Usual activities for 12 weeks followed by Moving Together classes (1 hour, 2 days/week) for 12 weeks.
- Moving Together - PLWD: Synchronous, online, mind-body group movement classes (1 hour, 2 days/week) for 12 weeks followed by return to usual activities for 12 weeks.
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 53
score on a scale | -1.7 (0.6) | 0.7 (4.2)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.048, Mixed Models Analysis; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [0.01 to 4.39] — The mean difference estimate of 2.2 was confirmed. It is slightly different than the difference of the raw change values [+.7 - (-1.7) = 2.4] because it comes from the mixed effects model

2. Primary Outcome: Caregiver Physical Health - Change (Short Form Health Survey [SF-12] Physical Composite Score [PCS])
Description: The Short Form Health Survey (SF-12) is a 12-item questionnaire that was developed as a shorter alternative to the SF-36 Health Survey (SF-36). It consists of a subset of 12 items from the SF-36 covering the same eight domains of health outcomes and generates two summary scores: the Physical and Mental Health Composite Scores (PCS, MCS). Scores may range from 0-100, with higher scores reflecting better levels of health.
Time Frame: Baseline to 12-weeks
Population: Measured only in CPs.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Waitlist Control - CP: Usual activities for 12 weeks followed by Moving Together classes (1 hour, 2 days/week) for 12 weeks.
- Moving Together - CP: Synchronous, online, mind-body group movement classes (1 hour, 2 days/week) for 12 weeks followed by return to usual activities for 12 weeks.
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 54 | 43
score on a scale | 0.2 (8.0) | -0.6 (7.7)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.603, Mixed Models Analysis; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-4.12 to 2.40]

3. Primary Outcome: Caregiver Mental Health - Change (Short Form - 12 [SF-12] Mental Composite Score [MCS])
Description: as for outcome 2
Time Frame: Baseline to 12 weeks
Population: Only measured in CPs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | -0.7 (7.9) | 0.0 (8.1)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.734, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.75 to 3.92]

4. Secondary Outcome: Well-being - Change (Neuro-QOL v1.0 Positive Affect and Well-Being Short Form)
Description: The Neuro-QOL v1.0 Positive Affect and Well-Being Short Form includes 9 items (e.g. sense of well-being, feeling hopeful, life was satisfying, etc.) with 5-point responses from never (1) to always (5). Scores range from 0-40 with higher scores indicating increased mobility.
Time Frame: Baseline to 12-weeks
Population: Only measured in PLWD. Data missing for 1 participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 53
score on a scale | -1.7 (6.1) | 0.1 (4.0)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.159, Mixed Models Analysis; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-0.62 to 3.74]

5. Secondary Outcome: Social Isolation - Change (Patient-Reported Outcomes Measurement Information System v2.0 Social Isolation Scale)
Description: The Patient-Reported Outcomes Measurement Information System v2.0 social isolation scale consists of 4 items (feeling left out, people barely know me, feeling isolated, people are around but not with me) that are rated as 1 (never), 2 (rarely), 3 (sometimes), 4 (usually), or 5 (always). Scores range from 0-20 with higher scores indicating less perceived social isolation.
Time Frame: Baseline to 12-weeks
Population: Measured in PLWD. Data missing for 1 participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 53
score on a scale | -0.2 (3.6) | -0.5 (4.4)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.818, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.97 to 1.56]

6. Secondary Outcome: Mobility - Change (Neuro-QOL Short Form V1.0 - Lower Extremity Function - Mobility)
Description: The (Neuro-QOL Short Form v1.0 -- Lower Extremity Function -- Mobility), which includes 8 items for functional mobility (getting on and off the toilet, getting in and out of a car, getting out of bed into a chair). Responses are rated on a 5-point Likert scale: 1( Without any difficult), 2 (With a little difficulty), 3 (With some difficulty), 4 (With much difficulty), 5 (Unable to do). Scores may range from 0-40 with higher scores indicating increased mobility.
Time Frame: Baseline to 12-weeks
Population: Measure applies to PLWD. Data missing for 1 Moving Together participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 53
score on a scale | -1.6 (5.0) | 0.3 (3.7)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.089, Mixed Models Analysis; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-0.26 to 3.51]

7. Secondary Outcome: Cognitive Function - Change (Telephone Montreal Cognitive Assessment, t-MoCA)
Description: The t-MoCA is extracted from the original face-to-face MoCA and uses items not requiring the use of a pencil and paper or visual stimulus. Scores may range from 0-22 with higher scores indicating higher cognitive function.
Time Frame: Baseline to 12-weeks
Population: Measured only in PLWD. Data missing for 1 Moving Together participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 53
score on a scale | -0.8 (3.3) | -0.5 (2.5)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.631, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.96 to 1.58]

8. Secondary Outcome: Caregiver Healthy Days - Change (Healthy Days Core Module)
Description: The Healthy Days Core Modules includes 3 questions about the number of days during the past 30 days that physical or mental health was not good or poor physical or mental health kept from doing usual activities. Scores range from 0-18 with lower scores indicating higher physical or mental health.
Time Frame: Baseline to 12-weeks
Population: Measure applies to CPs only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | 0.0 (2.5) | 0.5 (2.8)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.484, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.71 to 1.49]

9. Secondary Outcome: Caregiver Self-efficacy - Change (Gain in Alzheimer Care INstrument (GAIN))
Description: The GAIN consists of 10-items (e.g., increased my self-awareness, increased my knowledge and skills in dementia care) using a Likert scale from 0 (disagree a lot) to 4 (agree a lot). Scores range from 0 to 40 with higher scores indicating increased positive feelings about caregiving
Time Frame: Baseline to 12-weeks
Population: Measure applies to CPs only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | 0.1 (5.0) | 0.5 (7.4)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.81, Mixed Models Analysis; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.36 to 3.01]

10. Secondary Outcome: Caregiver Burden - Change (Zarit Burden Interview, 6-item Version)
Description: The Zarit Burden Interview is one of the most widely used assessments for caregiver burden covering areas including caregiver's health, psychological well-being, finances, social life, and the relationship between the caregiver and the person with dementia. Scores range from 0-24 with higher scores indicating positive caregiver experience.
Time Frame: Baseline to 12-weeks
Population: Measure applies to CPs only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | -0.2 (3.1) | 0.4 (3.5)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.384, Mixed Models Analysis; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.77 to 2.00]

11. Secondary Outcome: Caregiver Social Isolation - Change (PROMIS v2.0 Social Isolation Scale)
Description: as for outcome 5
Time Frame: Baseline to 12-weeks
Population: Measure applies to CPs only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | 0.3 (2.3) | -0.1 (3.4)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.509, Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.65 to 0.81]

12. Secondary Outcome: Caregiver Self-regulation - Change (Abbreviated Multidimensional Assessment of Interoceptive Awareness-2 (MAIA) Self-regulation Subscale)
Description: The MAIA-2 - Self-regulation subscale is designed to assess ability to regulate distress by attention to body sensations (e.g., when I feel overwhelmed, I can find a calm place inside). Scores range from 0-20 with higher scores indicating increased self-regulation.
Time Frame: Change from baseline to 12-weeks
Population: Measure applies to CPs only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | 0.3 (2.4) | 1.9 (3.9)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.021, Mixed Models Analysis; Mean Difference (Final Values) = 1.60, 95% CI 2-sided [0.24 to 3.01]

13. Secondary Outcome: Caregiver Positive Affect (Positive States of Mind)
Description: The Positive States of Mind scale is designed to assess types of positive mood (e.g., focused attention, productivity, responsible caregiving, etc.). This scale consists of 6-items using a 4-point Likert scale from 0 (Unable to have it) to 3 (Have it Easily). Scores range from 0-18 with higher scores indicating positive mood.
Time Frame: Baseline to 12-weeks
Population: Measure applies to CPs only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | 0.5 (2.1) | -0.3 (3.1)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.156, Mixed Models Analysis; Mean Difference (Final Values) = -0.80, 95% CI 2-sided [-1.94 to 0.31]

14. Secondary Outcome: Caregiver Sleep - Change (Symptom Checklist, 3 Items)
Description: The Symptom Checklist-90-Revised is a 90-item self-report questionnaire often used to assess global psychological distress and the investigators will be using 3 items assessing: trouble falling asleep, awakening in the early morning, and sleep that is restless or disturbed. Scores range from 0-12 with lower scores indicating less sleep difficulties.
Time Frame: Baseline to 12-weeks
Population: Measure only applies to CPs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 43 | 54
score on a scale | -0.1 (1.9) | 0.2 (2.1)
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.582, Mixed Models Analysis; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.62 to 1.10]

15. Secondary Outcome: People With Memory Loss (PWML) Sleep - Change (Symptom Checklist, 3 Items)
Description: Caregivers also will be asked about sleep for the PWML using the 3 sleep items from the Symptom Checklist-90-Revised (trouble falling asleep, awakening in the early morning, and sleep that is restless or disturbed). Scores range from 0-12 with lower scores indicating less sleep difficulties.
Time Frame: Baseline to 12-weeks
Population: Measure only asked of CPs regarding PLWD.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 54
score on a scale | 0.1 (2.0) | -0.3 (1.7)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.271, Mixed Models Analysis; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-1.21 to 0.34]

16. Secondary Outcome: People With Memory Loss (PWML) Mobility - Change (Neuro-QOL Short Form V1.0 - Lower Extremity Function - Mobility)
Description: As described above, the Neuro-QOL Short Form v1.0 - Lower Extremity Function - Mobility includes 8 items for functional mobility (e.g. getting on and off the toilet, getting in and out of a car, getting out of bed into a chair, etc.). CGs will be asked about the mobility of the PWML. Scores range from 0-35 with higher scores indicating less physical difficulty with daily activities.
Time Frame: Baseline to 12-weeks
Population: Measure asked of CPs regarding PLWD.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 54
score on a scale | -0.3 (4.9) | -0.2 (3.1)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.834, Mixed Models Analysis; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.52 to 1.88]

17. Secondary Outcome: People With Memory Loss (PWML) Cognitive Function - Change (Cognitive Function Instrument - Modified)
Description: The original Cognitive Function Instrument included 14 items that asked about decline in cognitive function (e.g., memory, tendency to repeat questions, misplacing things, etc.) compared to 1 year ago with responses of yes (1), no (0) or maybe (0.5). The investigators will be using a modified 11-item version that excludes items on driving, managing money, work; asking about change in the past 3 months (to match the duration of our study); and using a 5-point Likert scale from 1 (a lot worse) to 5 (a lot better). Scores range from 0-55 with higher scores indicating improved cognitive function.
Time Frame: Baseline to 12-weeks
Population: Measure asked CPs about PLWD.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 43 | 54
score on a scale | 1.5 (5.1) | 1.8 (6.1)
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.529, Mixed Models Analysis; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.62 to 3.15]

18. Other Pre Specified Outcome: Caregiver (CG) Falls
Description: Total number of falls reported for CG for the entire group (not per CG)
Time Frame: Baseline to 12 weeks
Population: Applies to CPs only. Data missing for 2 Waitlist and 6 Moving Together CPs.
Measure: Number; unit: falls
Arm/Group | Waitlist Control - CP | Moving Together - CP
Number analyzed (Participants) | 41 | 48
falls | 6 | 11
Statistical Analysis 1: Comparison: Waitlist Control - CP vs Moving Together - CP; Test type: Superiority; p = 0.377, Poisson regression

19. Other Pre Specified Outcome: People With Memory Loss (PWML) Falls
Description: Total number of falls reported for PWML in the entire group (not per participant).
Time Frame: Baseline to 12 weeks
Population: Applies only to PLWD. Data missing for 2 Waitlist and 6 Moving Together participants.
Measure: Number; unit: falls
Arm/Group | Waitlist Control - PLWD | Moving Together - PLWD
Number analyzed (Participants) | 41 | 48
falls | 26 | 16
Statistical Analysis 1: Comparison: Waitlist Control - PLWD vs Moving Together - PLWD; Test type: Superiority; p = 0.043, Poisson regression

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Care partners are sent a month survey that asks about hospitalizations, emergency department visits, falls, and other unexpected major medical events or changes to health in the past month for themselves and PLWD. We did not group events by organ system; therefore, they are reported as general events.
Groups:
- Immediate Start - Care Partners (CPs); Immediate Start - Participants Living With Dementia (PLWD): The Immediate Start group will participate in Moving Together classes (1 hour, 2 days/week) for 12 weeks and will then return to usual activities for 12 weeks. Adverse events are reported separately for care partners (CPs) and participants living with dementia (PLWD).
- Delayed Start - Care Partners (CPs); Delayed Start - Participants Living With Dementia (PLWD): The Delayed Start group will engage in usual activities for 12 weeks and will then participate in Moving Together classes (1 hour, 2 days/week) for 12 weeks. Adverse events are reported separately for care partners (CPs) and participants living with dementia (PLWD).
Arm/Group | Immediate Start - Care Partners (CPs) | Immediate Start - Participants Living With Dementia (PLWD) | Delayed Start - Care Partners (CPs) | Delayed Start - Participants Living With Dementia (PLWD)
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/54 | 7/54 | 1/43 | 3/43
Other Adverse Events (participants affected / at risk) | 3/54 | 17/54 | 8/43 | 15/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start - Care Partners (CPs) (N=54) | Immediate Start - Participants Living With Dementia (PLWD) (N=54) | Delayed Start - Care Partners (CPs) (N=43) | Delayed Start - Participants Living With Dementia (PLWD) (N=43)
Other (General disorders) | 1 (1) | 7 (11) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Start - Care Partners (CPs) (N=54) | Immediate Start - Participants Living With Dementia (PLWD) (N=54) | Delayed Start - Care Partners (CPs) (N=43) | Delayed Start - Participants Living With Dementia (PLWD) (N=43)
Any Adverse Event (General disorders) | 3 (10) | 17 (32) | 8 (14) | 15 (34)

LIMITATIONS AND CAVEATS:
Dyads were enrolled in cohorts with a goal of 16 dyads per cohort. Our original target sample size of 224 dyads (112/group) was reduced to 112 dyads (56/group) following a futility analysis requested by our Safety Officer (SO). We did not penalize the alpha for this unplanned interim analysis. Due to time and funding constraints, the 7th (final) cohort only included 10 dyads, all of whom were assigned to the Immediate Start (Moving Together) group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT04621448/Prot_SAP_000.pdf